CLINICAL TRIAL: NCT05132387
Title: Wroclaw Out-Of-Hospital Cardiac Arrest Registry
Acronym: WOHCA
Status: Recruiting | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Collaborators: Wroclaw Emergency Medical Services (Unknown)
Responsible Party: Principal Investigator, Wiktor Kuliczkowski, Head of the Cardiac Catheterisation Laboratory, Wroclaw Medical University
Other Study IDs: 327/2021
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Cardiac arrest, ECMO, ECMO-CPR
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Out-of-hospital cardiac arrest: Patients with out-of-hospital cardiac arrest which occured in the predefined area of the city of Wroclaw.
  Interventions: Other: ECMO assisted CPR in out-of-hospital cardiac arrest

INTERVENTIONS:
Other: ECMO assisted CPR in out-of-hospital cardiac arrest — Patients included in the registry will be transferred during LUCAS assisted CPR by the Wroclaw Emergency Medical Services to the Emergency Department of the Wroclaw University Hospital where blood gasses will be assessed. If two or more of the following: end-tidal carbon dioxide (CO2) > 10 mm Hg, arterial partial pressure of oxygen (PaO2) >50 mm Hg or oxygen saturation >85%, and lactic acid <18 mmol/L will be fulfilled patient will be further transferred to the Cardiac Catheterization Laboratory for V-A ECMO implantation followed by coronary/pulmonary artery angiography and intervention.

SUMMARY:
The purpose of this study is to assess the efficacy of institutionalized care program of patients with out-of-hospital cardiac arrest.

DETAILED DESCRIPTION:
Patients with out-of-hospital cardiac arrest included in the program will be treated with extracorporeal membrane oxygenation (ECMO) assisted cardiopulmonary resuscitation (CPR) with additional invasive procedures including coronary/pulmonary angiography and intervention. This type of treatment was not provided in institutionalized fashion in Wroclaw, Poland. Implementation of this program should improve survival in out-of-hospital cardiac arrest patients, which currently is less than 10%.

ELIGIBILITY:
Inclusion Criteria:

* Age < 60 years
* witnessed sudden cardiac arrest with immediate CPR
* supposed cardiac cause of the event
* ventricular fibrillation (VF) or pulseless ventricular tachycardia (VT) at first medical contact with 3 unsuccessful defibrillations (no ROSC)
* CPR conducted with Lund University Cardiopulmonary Assist System (LUCAS™)
* Estimated transfer time from the scene to the Emergency Department < 30 minutes.
* End tidal carbon dioxide (ETCO2) > 10 mmHg

Exclusion Criteria:

* Total presumed time from 112 call to ECMO implantation longer than 60 minutes
* Age < 18 years old or > 60 years old;
* Non-shockable initial rhythm
* Unavailability of the automated CPR device
* Unavailability of the catheterisation laboratory
* Severe concomitant illness with decreased life expectancy
* Severe body injury
* Severe active bleeding
* Drowning
* Terminal cancer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with out-of-hospital cardiac arrest which occured in the predefined area of the city of Wroclaw, Poland.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 1 month
  all cause mortality

SECONDARY OUTCOMES:
degree of disability | 3 and 6 months after index event
  Modified Rankin Scale of 3 or lower

CONTACTS AND LOCATIONS:
Overall Officials: Wiktor Kuliczkowski, MD, Principal Investigator — Wroclaw Medical University
Locations (1):
- Wroclaw University Hostpital, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sip M, Puslecki M, Klosiewicz T, Zalewski R, Dabrowski M, Ligowski M, Goszczynska E, Paprocki C, Grygier M, Lesiak M, Jemielity M, Perek B. A concept for the development of a pioneer regional Out-of-Hospital Cardiac Arrest Program to improve patient outcomes. Kardiol Pol. 2020 Sep 25;78(9):875-881. doi: 10.33963/KP.15433. Epub 2020 Jun 16. PMID 32550730
- [Background] Yannopoulos D, Bartos J, Raveendran G, Walser E, Connett J, Murray TA, Collins G, Zhang L, Kalra R, Kosmopoulos M, John R, Shaffer A, Frascone RJ, Wesley K, Conterato M, Biros M, Tolar J, Aufderheide TP. Advanced reperfusion strategies for patients with out-of-hospital cardiac arrest and refractory ventricular fibrillation (ARREST): a phase 2, single centre, open-label, randomised controlled trial. Lancet. 2020 Dec 5;396(10265):1807-1816. doi: 10.1016/S0140-6736(20)32338-2. Epub 2020 Nov 13. PMID 33197396